CLINICAL TRIAL: NCT03180606
Title: Enhanced Primary Care for Elderly: A Multicenter Pragmatic Clinical Trial Where Older People With Great Needs Are Predicted and Given Personalized Primary Care
Brief Title: Enhanced Primary Care for Elderly
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Jan Marcusson, MD, senior consultant, professor, Region Östergötland
Other Study IDs: Elderly care 2016-347-31
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Frail Elderly Syndrome
Keywords: Elderly; Frail; Primary care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Predicted and personalized primary care: Elderly 75 years of age and older in primary care with high risk of being fragile and future risk of needing hospital care that receives personalized primary care
  Interventions: Other: Multi-disciplinary and personalized primary care
- Predicted but with treatment as usual: Elderly 75 years of age and older in primary care with high risk of being fragile and future risk of needing hospital care that receives treatment as usual

INTERVENTIONS:
Other: Multi-disciplinary and personalized primary care — Team-based primary care where nurse, GP, social-worker, physiotherapist, occupational therapist evaluate and give treatment
  Groups: Predicted and personalized primary care

SUMMARY:
The present health care situation for the elderly in many countries is insufficient and not designed according to the health care needs of the aged population. In a pragmatic multicenter primary care setting (n= 1600), the investigators use an evidence based prediction model to find elderly (75+) with high risk for complex medical care or hospitalization and apply a differentiated and directed medical and social care to this risk group, in comparison to usual care. The intervention will include all the latest evidence based tools in the care of elderly (multi-professional team, social support, medical care home-visits, telephone support, general practitioner visits, etc). The project has high potential impact on the development of future care of elderly.

In addition to the intervention study, several academic sub-studies focusing on patient's perspective, professional roles, equality, implementation and governance management of health care will be performed.

DETAILED DESCRIPTION:
The current project is a multidisciplinary research project covering several aspects of a shift in elderly care, with outcome measures not only related to primary medical or functional measures. The analyses will widen the view to overall societal costs and effects of changes in key institutions of social security as well as to hidden mechanisms in the governance system of care and health care of elderly.

The primary aim of the present study is to investigate the extent to which a differentiated (personalized) and targeted primary care intervention provided to a statistically predicted risk population of elderly, results in care that is more effective and of higher quality than that of a control group receiving standard care. In a pragmatic multicenter primary care setting (n= 1600), an evidence based prediction model to find elderly (75+) with high risk for complex medical care or hospitalization is used followed by a differentiated and directed medical and social care to this risk group, in comparison to usual care. The intervention will include all the latest evidence based tools in the care of elderly (multi-professional team, social support, medical care home-visits, telephone support, general practitioner visits, etc).

The investigators also aim to study the care model in a broader sense; experiences of the elderly, their social networks and diversity. Finally, the project will also investigate how the health care system, from specific health care professionals (primary care nurses, doctors, para-medical staff) to management levels and politicians influence the implementation of the present and future care models. One specific subproject focuses on the mechanisms behind the inability of steak holders/politicians and top administrative executives to find efficient governance principals for elderly care and health care, despite already available knowledge sources.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and older living in county of Östergötland

Exclusion Criteria:

* No exclusion criteria

Ages: 75 Years to 110 Years | Sex: All
Age Groups: Older Adult
Study Population: People 75 years and older in the county of Östergötland with a high risk of being fragile and in need of hospital care. This risk group of 1600 out of 24000 is detected by a digital/statistical method depending on previous health care consumption and specific diagnoses
Sampling Method: Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital care days | January 1st 2018 - December 31st 2019
  The number of days in hospital

SECONDARY OUTCOMES:
Hospital care occasions | January 1st 2018 - December 31st 2019
  Number of occasions in hospital care
Health related quality of life | January 1st 2018 - December 31st 2019
  Measured as EQ-5D scores
Costs for health care | January 1st 2018 - December 31st 2019
  The total costs for health care measured in USD
Mortality | January 1st 2018 - December 31st 2019
  Number of deaths during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Jan Marcusson, MD, PhD, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Region Östergötland/Linköping University, Linköping, Östergötland County
  - Primary Care of Östergötland, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marcusson J, Nord M, Johansson MM, Alwin J, Levin LA, Dannapfel P, Thomas K, Poksinska B, Sverker A, Olaison A, Cedersund E, Kelfve S, Motel-Klingebiel A, Hellstrom I, Kullberg A, Bottiger Y, Dong HJ, Peolsson A, Wass M, Lyth J, Andersson A. Proactive healthcare for frail elderly persons: study protocol for a prospective controlled primary care intervention in Sweden. BMJ Open. 2019 May 22;9(5):e027847. doi: 10.1136/bmjopen-2018-027847. PMID 31122995
- [Derived] Hansen K, Lyth J, Segernas A, Alwin J, Nord M. Self-rated health as a predictor of mortality and healthcare use in older adults at high risk of hospitalisation: a prospective cohort study in Sweden. BMJ Open. 2025 Sep 1;15(9):e091787. doi: 10.1136/bmjopen-2024-091787. PMID 40889980
- [Derived] Dong HJ, Yang J, Johansson MM, Peolsson A, Barbero M, Nord M. Association between frailty and pain in older people at high risk of future hospitalization. Front Pain Res (Lausanne). 2025 Apr 28;6:1576691. doi: 10.3389/fpain.2025.1576691. eCollection 2025. PMID 40386744
- [Derived] Dong HJ, Peolsson A, Johansson MM. Effects of proactive healthcare on pain, physical and activities of daily living functioning in vulnerable older adults with chronic pain: a pragmatic clinical trial with one- and two-year follow-up. Eur Geriatr Med. 2024 Jun;15(3):709-718. doi: 10.1007/s41999-024-00952-9. Epub 2024 Mar 6. PMID 38446408
- [Derived] Lundgren M, Segernas A, Nord M, Alwin J, Lyth J. Reasons for hospitalisation and cumulative mortality in people, 75 years or older, at high risk of hospital admission: a prospective study. BMC Geriatr. 2024 Feb 20;24(1):176. doi: 10.1186/s12877-024-04771-2. PMID 38378482
- [Derived] Kammerlind AS, Peolsson A, Johansson MM. Dizziness in older persons at high risk of future hospitalization: prevalence, differences between those with and without dizziness, and effect of a proactive primary care intervention. BMC Geriatr. 2022 Apr 10;22(1):315. doi: 10.1186/s12877-022-02910-1. PMID 35399055
- [Derived] Nord M, Lyth J, Alwin J, Marcusson J. Costs and effects of comprehensive geriatric assessment in primary care for older adults with high risk for hospitalisation. BMC Geriatr. 2021 Apr 21;21(1):263. doi: 10.1186/s12877-021-02166-1. PMID 33882862
- See also: Study protocol article — http://dx.doi.org.e.bibl.liu.se/10.1136/bmjopen-2018-027847